CLINICAL TRIAL: NCT04275375
Title: Department of Anaesthesiology, Taipei Veterans General Hospita, Taipei, Taiwan
Brief Title: Autonomic Modulation After Spinal Anesthesia With Depth of Anesthesia and Vital Signs.
Status: Completed | Type: Observational
Sponsor: National Central University (Other)
Responsible Party: Principal Investigator, Hsin-Yi Wang, Principal Investigator, National Central University
Other Study IDs: 2019-01-016CC
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Participants Scheduled for Surgery Under Spinal Anesthesia Without Impairment of Renal, Hepatic, Cardiac or Respiratory Function
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- hyperbaric bupivacaine: The dosage of hyperbaric bupivacaine decided by the clinical anesthesiologist. This study is an observational study.
  Interventions: Other: observation study about the autonomic response after spinal anesthesia
- plain bupivacaine: The dosage of plain bupivacaine decided by the clinical anesthesiologist. This study is an observational study.
  Interventions: Other: observation study about the autonomic response after spinal anesthesia

INTERVENTIONS:
Other: observation study about the autonomic response after spinal anesthesia — ECG waveforms were continuously recorded using a multichannel polygraphic system (Embla N7000, Natus, Pleasanton, CA). The data were saved at a rate of 1024 Hz directly to a memory card within the device for offline analysis of heart rate variability (HRV) and PPG. All data included in the analysis were obtained from continuous artifact-free ECG recordings for analysis of the immediate effects of spinal anesthesia.

SUMMARY:
Spinal anaesthesia has the advantage that produced nerve block by the injection of local anaesthetic into cerebrospinal fluid (CSF). However, the greatest challenge in spinal anaesthesia is to control the spread of local anaesthetic through the CSF to provide a block which is adequate for the proposed surgery without unnecessary extensive spread, and increased risk of complications.

DETAILED DESCRIPTION:
The activity of the autonomic nervous system is of fundamental importance in the regulation of vital bodily functions. Unbalance of autonomic nerve system results in considerably disordered vital function. Clinically, this is of great significance, because if an anesthetic agent produces cause the sympathetic system to block, the effects can be serious in individual cases, particularly on the cardiovascular system. If complications are to be avoided, it is essential to assess the degree of block correctly. Clinical monitoring has a variety of applications, a particularly useful one being measurement of the sympathetic system during regional anesthesia, for which quantification of the blocking effect is a clinical necessity and the degree of block needs to be ascertained without delay. The autonomic nervous system (ANS) plays an important role in the regulation of hemodynamics during anesthesia. Analysis of beat-to-beat fluctuations of heart rate and blood pressure is a promising new approach to the clinical diagnosis and management of alterations in cardiovascular regulation. Continuous Wavelet Transform (CWT), which could overcome the limitation of the steady-state assumption in the classical spectral analysis, is believed as a reliable and robust method to access cardiorespiratory dynamics of the ANS and the investigators will applied during spinal anesthesia to evaluate the detail changes.

ELIGIBILITY:
Inclusion Criteria:

1. patients scheduled for operation with spinal anesthesia

Exclusion Criteria:

1. recently treat with a sedative, beta-blocker, parasympatholytic, or opioid agent
2. emergency surgery
3. hypovolemia and hypothermia, arrhythmia, diabetes, or impairment of renal, hepatic, coagulation, cardiac, or respiratory function

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators conducted a prospective observational study on patients who were scheduled to undergo elective surgery and spinal anesthesia. The investigators excluded patients who had recently been treated with a sedative, beta-blocker, parasympatholytic, or opioid agent, patients who had undergone emergency surgery, those with hypovolemia and hypothermia, arrhythmia, diabetes, or impairment of renal, hepatic, coagulation, cardiac, or respiratory function
Sampling Method: Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2019-03-01 (Actual); Primary Completion 2019-08-16 (Actual); Study Completion 2019-08-16 (Actual)

PRIMARY OUTCOMES:
record and compare changes in ANS function( HRV and PPGA) after spinal anesthesia in different group | maximum for 4 hours
  Electrocardiography and pulse photoplethysmography signals were recorded after spinal anesthesia. The spectrogram of beat-to-beat R-to-R intervals was derived by continuous wavelet transform (CWT), and the immediate power of high frequency (HFi) and low frequency (LFi) bands was extracted at
  1-second intervals. The derived parameters, HF, LF, and pulse photoplethysmography amplitude, were normalized by their maximum and minimum values. Mixed-model regression and repeated-measures analysis of variance were used to explore the time-dependent effect.

CONTACTS AND LOCATIONS:
Locations (1):
- Taipei Veterans General Hospital, Taipei, R.o.c, Taiwan